CLINICAL TRIAL: NCT02356549
Title: African American Cancer Clinical Trial Decisions: Testing Tailored Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: MCC-14-10762; HM20002965 (Other: Virginia Commonwealth University); NCI-2015-01819 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2015-01-15; First posted 2015-02-05 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Myeloma; Lymphoma; Leukemia
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma; Leukemia | interventions — Electronic Health Records

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP 1: (EMR) Tailoring Alone (Active Comparator): Patients will be randomized to receive tailored messages based on demographic and disease information extracted from Massey Cancer Center (MCC) electronic medical records (EMR) that will include a) demographic information: age, income, education and health insurance status, b) disease variables: cancer type and severity and c) trial variables: phase of trial being offered and prior trial participation.
  Interventions: Behavioral: EMR Tailoring
- GROUP 2:EMR Tailoring+Feedback (Active Comparator): Patients will be randomized to receive tailored messages based on information extracted from the EMR as in Group 1. Physicians also receive a summary of tailored messages provided to patients.
  Interventions: Behavioral: EMR Tailoring; Behavioral: Physician Involvement
- GROUP 3:EMR+Survey Tailoring alone (Active Comparator): Patients will be randomized to receive tailored messages based on EMR data as in Group 1. Patients will complete a survey that will be used to provide a deeper level of tailored messages
  Interventions: Behavioral: EMR Tailoring; Behavioral: Survey Tailoring
- GROUP 4:EMR+Survey Tailoring+Feedback (Active Comparator): Patients will be randomized to receive tailored messages based on information extracted from their EMR as in Group I. Patients will complete a survey that will be used to provide a deeper level of tailored messages as in Group 3. Physicians also receive a summary of tailored messages provided to patients as in Group 2.
  Interventions: Behavioral: EMR Tailoring; Behavioral: Survey Tailoring; Behavioral: Physician Involvement

INTERVENTIONS:
Behavioral: EMR Tailoring — Electronic Medical Records (EMR) data alone will be entered into the Michigan Tailoring System (MTS system) and their brochures will be prepared.
  Other Names: "shallow" level of tailored messages; EMR; Electronic Medical Records (EMR) Tailoring
Behavioral: Survey Tailoring — Survey that will use standardized, psycho-metrically sound measures to gather information about patients, including their levels of trust in medical research and preferences for information and decision involvement. The survey augmented by their EMR data will be used to develop a level of tailored messages.
  Other Names: "deeper" level of tailored messages; Tailoring Survey; deep tailoring; Survey data tailoring
  Arms: GROUP 3:EMR+Survey Tailoring alone; GROUP 4:EMR+Survey Tailoring+Feedback
Behavioral: Physician Involvement — Prior to the consultation, physicians of patients will receive a summary of patients' tailored message brochure from the Research Assistant (RA) and included in the patient's notes. At the conclusion of the consultation, the RA will ask the oncologist whether or not a clinical trial was discussed and whether or not they read the patients brochure.
  Other Names: Feedback
  Arms: GROUP 2:EMR Tailoring+Feedback; GROUP 4:EMR+Survey Tailoring+Feedback

SUMMARY:
The purpose of this study is to determine if the use of tailored health messages and/or involving physicians are effective in increasing African American (AA) patient activation in a clinical trial consultation. The proposal will use a composite score for patient activation derived from the Street Patient Activation Coding system. This will help to determine the effectiveness of our intervention on patient activation and patient centered clinical trial decision.

DETAILED DESCRIPTION:
A randomized clinical trial (using a 2x2 factorial design) to inform our knowledge of the efficacy of a tailored health message intervention, using different depths of tailoring and involving physicians, on AA cancer patients' active communication in CT consultations as measured by the Street Patient Activation measure. In this study 357 AA cancer patients will be randomized into one of four experimental groups Group 1 - messages tailored on Electronic Medical Record (EMR) data. Group 2 - messages tailored on EMR + physician involvement. Group 3 - messages tailored on EMR + survey. Group 4 - Messages tailored on EMR + survey + physician involvement. We will also measure patient: a) trust in their physician, b) trust in medical research, c) preferences that include information and decision involvement, d) communication self-efficacy, e) patient-family member communication congruence, f) consultation satisfaction and g) decision outcomes that include decisional conflict, decision satisfaction and decision regret.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age or older
* Have a cancer diagnosis
* Self identify as African American
* Therapeutic Phase I, II or III clinical trial at Massey Cancer Center (regardless of whether or not they join the therapeutic trial)
* Be able to provide informed consent
* We will also recruit one family member/caregiver (N = 357) of each participating patient
* Consented patients will not be excluded from this study if their family member declines to participate by completing the Cancer Communication Assessment Tool for Families (CCAT-F).

Exclusions Criteria:

-None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate the efficacy of the tailored health message intervention to increase patient activation. | 40 days
  Randomized clinical trial (using a 2x2 factorial design) to inform our knowledge of the efficacy of a tailored health message intervention, using different depths of tailoring and involving physicians, on AA cancer patients' active communication in CT consultations. In this study AA cancer patients will be randomized into one of four experimental groups. Scientifically determine the effectiveness of our intervention by using a composite score for patient activation derived from the Street Patient Activation Coding system.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brown, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Brown RF, Davis R, Wilson Genderson M, Grant S, Cadet D, Lessard M, Alpert J, Ward J, Ginder G. African-American patients with cancer Talking About Clinical Trials (TACT) with oncologists during consultations: evaluating the efficacy of tailored health messages in a randomised controlled trial-the TACT study protocol. BMJ Open. 2016 Dec 16;6(12):e012864. doi: 10.1136/bmjopen-2016-012864. PMID 27986738